CLINICAL TRIAL: NCT06018857
Title: Registry 17-009: Multi-Institutional Study Examining Patients With HCC Undergoing Liver Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Federico Aucejo (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Federico Aucejo, Director Liver Cancer Program, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 17-009
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a registry study examining patients with HCC undergoing liver transplantation including outcomes and predictors of recurrence

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age>18 years) undergoing Liver transplant for hepatocellular carcinoma

Exclusion Criteria:

* Patients under 18 years old
* Patients who do not have hepatocellular carcinoma
* patients who have hepatocellular carcinoma but do not undergo liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age>18 years) undergoing Liver transplant for hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | From date of surgery to date of identified cancer recurrence through either clinical judgement or scans. This is assessed up to 10 years after the surgery.
Overall Survival | From date of surgery to date of death, up to 10 years after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Aucejo, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wehrle CJ, Raj R, Maspero M, Satish S, Eghtesad B, Pita A, Kim J, Khalil M, Calderon E, Orabi D, Zervos B, Modaresi Esfeh J, Whitsett Linganna M, Diago-Uso T, Fujiki M, Quintini C, Kwon CD, Miller C, Pinna A, Aucejo F, Hashimoto K, Schlegel A. Risk assessment in liver transplantation for hepatocellular carcinoma: long-term follow-up of a two-centre experience. Int J Surg. 2024 May 1;110(5):2818-2831. doi: 10.1097/JS9.0000000000001104. PMID 38241354